CLINICAL TRIAL: NCT03475459
Title: A Clinical Pharmacology Study of NPC-15 to Evaluate Arrhythmogenic Effect in Healthy Adults
Brief Title: Investigation of Arrhythmogenic Effect of NPC-15 (NPC-15-7)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nobelpharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC-15-7
Record Dates: First submitted 2018-02-22; First posted 2018-03-23 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-04

CONDITIONS: Qt Interval, Variation in
Keywords: QTc prolongation effect

STUDY DESIGN:
Masking Description: This study is a single-arm, open label, dose escalation study. QT interval will be evaluated by blinding outcome assessor in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study drug (Experimental): Study drug (NPC-15 and/or Placebo ) will be orally administered once with 200 ml of water at 20:00 on the first days of Period I, Period II and Period III.
  Interventions: Drug: NPC-15 and/or Placebo

INTERVENTIONS:
Drug: NPC-15 and/or Placebo — The dosage and regimen of the study drug in each period is the following. Period I : NPC-15 placebo granules 8 g Period II : NPC-15 placebo granules 4 g + NPC-15 granules 0.2% 4 g (melatonin 8 mg) Period III : NPC-15 granules 0.2% 8 g (melatonin 16 mg)
  Other Names: Melatonin and/or Placebo

SUMMARY:
A study to assess the QTc prolongation effect of NPC-15 (melatonin 8mg or 16mg)

DETAILED DESCRIPTION:
This study is a single center, open label, dose escalation trial to evaluate prolongation effect on QT interval of NPC-15 (melatonin 8mg or 16mg).

The trial compose of 3 periods; During the each period, eligible volunteers wll be administered placebo, NPC-15 4g (melatonin 8mg) and NPC-15 8g(melatonin 16mg) as a sequential manner.

ELIGIBILITY:
Inclusion Criteria:

* Subject with BMI ≥ 17.6 kg/m2 and < 30.0 kg/m2.
* Subject who falls asleep at between 21:00 and 25:00 and wakes up at between 5:00 and 9:00 during 1 week prior to the first study drug administration.
* Subject who is able to comply with the study requirements during the study period.

Exclusion Criteria:

* Subject with QTcF interval greater than 450 ms in male or greater than 470 ms in female on the 12-lead electrocardiogram (ECG), or with clinically significant ECG abnormalities in other findings.
* Subject who has a family history of Torsades de Pointes (TdP) or long QT syndrome.
* Subject who has a history of hypersensitivity or allergies to melatonin or ramelteon.
* Subject who has a current or a history of disease which is considered inappropriate to be involved in the study, or who has any current disease to require treatments.
* Subject who received any non-prescription or prescription drug within 2 weeks prior to the first study drug administration.
* Subject who received any product containing St Jones Wart or any supplement containing melatonin within 4 weeks prior to the first study drug administration.
* Subject who has a history of smoking habit or was possibly exposed to passive smoking on a daily basis within 24 weeks prior to the first study drug administration.
* Subject who, in the opinion of the investigator or sub-investigator, is unsuitable to be involved in the study.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2018-04-29 (Actual); Study Completion 2018-04-29 (Actual)

PRIMARY OUTCOMES:
Time matched, baseline-adjusted change in Fridericia-corrected QTc (QTcF) intervals | Day1 and Day2 of each periods (3 periods)
  QTcF interval is a common endpoints to evaluate arrhythmogenic effect of test drug

SECONDARY OUTCOMES:
Serum melatonin concentration | Up to 12 hours post dose in each period (3 periods)
  NPC-15 is a preparation containing melatonin , therefore the change in blood concentration of melatonin is useful to evaluate the QTc prolongation effect of NPC-15.
Maximum drug concentration (Cmax) of melatonin | Up to 12 hours post dose in each period (3 periods)
  NPC-15 is a preparation containing melatonin , therefore pharmacokinetic parameter is useful to evaluate the QTc prolongation effect of NPC-15.
Maximum drug concentration time (Tmax) of melatonin | Up to 12 hours post dose in each period (3 periods)
  NPC-15 is a preparation containing melatonin , therefore pharmacokinetic parameter is useful to evaluate the QTc prolongation effect of NPC-15.
Area under the blood concentration time curve (AUC) of melatonin | Up to 12 hours postdose in each period (3 periods)
  NPC-15 is a preparation containing melatonin , therefore pharmacokinetic parameter is useful to evaluate the QTc prolongation effect of NPC-15.
Terminal elimination rate constant (λz) of melatonin | Up to 12 hours post dose in each period (3 periods)
  NPC-15 is a preparation containing melatonin , therefore pharmacokinetic parameter is useful to evaluate the QTc prolongation effect of NPC-15.
Mean residence time (MRT) of melatonin | Up to 12 hours postdose in each period (3 periods)
  NPC-15 is a preparation containing melatonin , therefore pharmacokinetic parameter is useful to evaluate the QTc prolongation effect of NPC-15.
Elimination half-life (t1/2) of melatonin | Up to 12 hours post dose in each period
  NPC-15 is a preparation containing melatonin , therefore pharmacokinetic parameter is useful to evaluate the QTc prolongation effect of NPC-15.
Clearance (CL) of melatonin | Up to 12 hours post dose in each period (3 periods)
  NPC-15 is a preparation containing melatonin , therefore pharmacokinetic parameter is useful to evaluate the QTc prolongation effect of NPC-15.
Volume of distribution (Vd) of melatonin | Up to 12 hours postdose in each period (3 periods)
  NPC-15 is a preparation containing melatonin , therefore pharmacokinetic parameter is useful to evaluate the QTc prolongation effect of NPC-15.
Adverse Events | Up to 36 hours post dose of Period III
  All events that emerge during treatment, having been absent pretreatment, or worsens relative to the pretreatment state

CONTACTS AND LOCATIONS:
Overall Officials: Masaharu Hayashi, MD, PhD, Principal Investigator — Shukutoku University
Locations (1):
- SOUSEIKAI Hakata Clinic, Fukuoka, Japan